CLINICAL TRIAL: NCT04450732
Title: A Phase 1, First-In-Human, Multicenter, Open-Label, Study of GQ1001, a HER2 Targeted Antibody-Drug Conjugate, Administered Intravenously, in Adult Patients With HER2-Positive Advanced Solid Tumors
Brief Title: Safety of GQ1001 in Adult Patients With HER2-Positive Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GeneQuantum Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GQ1001X2101
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: HER2-positive Breast Cancer; HER2-positive Biliary Tract Cancer; HER2-Positive Salivary Gland Carcinomas; HER2-Positive Advanced Solid Tumor
Keywords: HER2-positive; Biliary Tract Cancer; Salivary Gland Carcinomas; Non- Small Cell Lung Cancer; Advanced Solid Tumor
MeSH Terms: conditions — Biliary Tract Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Modified 3+3 Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): GQ1001 will be administered intravenously every 21 days. Dose Escalation will be guided by a modified 3+3 design.
  Interventions: Drug: GQ1001
- Dose Expansion (Experimental): GQ1001 at the Dose Recommended for Dose Expansion will be administered intravenously every 21 days. Dose expansion will further evaluate the MTD or DRDE in different types of malignant solid tumor in four cohorts.
  Interventions: Drug: GQ1001

INTERVENTIONS:
Drug: GQ1001 — anti-HER2 antibody drug conjugate

SUMMARY:
Phase I Dose Finding Study for GQ1001 in Patients with HER2-Positive Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form and able to comply with the protocol;
2. Male and female subjects ≥18 years of age;
3. ECOG PS of 0 or 1, the estimated life expectancy ≥ 3 months;
4. LVEF ≥ 50% as determined by echocardiography (ECHO);
5. Patients must have pathologically documented advanced/unresectable or metastatic solid tumor with HER2-positive (as defined below) that is relapsed or refractory to standard therapy or for which there is no standard therapy and progressed. Patients must have a least one measurable disease lesion. Tumor specimens to identify HER2 status should be obtained within the past 6 months.

   Definition of HER2-positive
   * Advanced/unresectable or metastatic breast cancer: immunohistochemistry (IHC) 3+, or IHC 2+ and in situ hybridization positive (ISH+)*;
   * Advanced/unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma: IHC 3+, or IHC 2+ and ISH+*;
   * Other HER2-positive advanced/unresectable or metastatic solid malignant tumor: determined by IHC, ISH, Next Generation Sequencing, or other analysis techniques as appropriate;

     * ISH: fluorescence in situ hybridization (FISH) or dual in situ hybridization (DISH); ISH positivity is defined as a ratio of ≥ 2.0 for the number of HER2 gene copies to the number of signals for CEP17. ISH assay is not required when IHC result is 3+. ISH assay should be performed to confirm HER2 positivity when IHC result is 2+.
6. Adequate organ function confirmed at screening and within 7 days before the first treatment, as evidenced by:

   Platelet count: ≥ 100,000/mm3 ; Hemoglobin : ≥ 9 g/dL; Absolute neutrophil count (ANC): ≥ 1500/mm3 ; Serum creatinine: ≤ 1.5 × ULN (upper limit of normal), or creatinine clearance ≥ 60 mL/min (using Cockcroft Gault formula) ; Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) : ≤ 2.5 × ULN (≤ 5 × ULN if liver metastases are present); Total bilirubin : ≤ 1.5 × ULN (except for patients with Gilbert's Syndrome); Prothrombin time and activated partial thromboplastin time: ≤ 1.5 × ULN.
7. Adequate washout period before the first treatment as defined by:

   Major surgery: ≥ 4 weeks. Radiation therapy: ≥ 4 weeks (≥ 2 weeks for palliative stereotactic radiation therapy without abdominal). Autologous transplantation: ≥ 3 months.

   Hormonal therapy: ≥ 2 weeks or per Investigator's discretion for breast cancer patients.

   Chemotherapy or targeted therapy (including antibody drug therapy): ≥ 3 weeks (≥ 2 weeks for 5 flourouracil-based agents, folinate agents, and/or weekly paclitaxel; ≥ 2 weeks (or 5 half-lives, whichever is shorter) for tyrosine kinase inhibitors; ≥ 4 weeks for HER2-directed biologic therapies; ≥ 6 weeks for nitrosoureas or mitomycin C). Immunotherapy: ≥ 4 weeks. Strong cytochrome P450 enzyme 3A4 (CYP3A4) inhibitor: ≥ 3 elimination half-lives . Any investigational agents or treatments: ≥ 4 weeks.
8. Patients without a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections or with a history of AIDS-defining opportunistic infections and have not had an opportunistic infection within the past 12 months may be enrolled per the discretion of the Investigator.

Exclusion Criteria:

1. Clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of chemotherapy or radiotherapy;
2. Subjects with multiple primary malignancies within 2 years, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, other solid tumors curatively treated, or contralateral breast cancer);
3. Cardiovascular dysfunction or clinically significant cardiac disease, including but not limited to:

   * Medical history of symptomatic chronic heart failure (New York Heart Association (NYHA) classes II-IV) or serious cardiac arrhythmia requiring treatment;
   * Medical history of myocardial infarction or unstable angina within 6 months of the first treatment;
   * Corrected QT interval by Fridericia (QTcF) prolongation of > 450 milliseconds (ms) in males and > 470 ms in females;
4. Medical history of clinically significant lung disease (e.g., interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis), or patients who are suspected to have these diseases by imaging at screening or requirement for supplemental oxygen;
5. Known hypersensitivity to either the drug substances or inactive ingredients in the drug product;
6. Existing Grade ≥ 2 peripheral neuropathy;
7. Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI CTCAE version 5.0, Grade ≤ 1 or baseline. Subjects with chronic Grade 2 toxicities may be eligible per the discretion of the Investigator;
8. Cumulative anthracycline dose > 360 mg/m2 doxorubicin or equivalent;
9. Uncontrolled infection requiring i.v. of antibiotics, antivirals or antifungals;
10. Active infection with hepatitis C (e.g., detectable antibodies to hepatitis C virus [HCV]) or hepatitis B (e.g., hepatitis B surface antigen [HBsAg] positive) except subjects with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative HBsAg) may be included if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is undetectable at the time of screening, and these subjects must be willing to undergo monthly DNA testing and appropriate antiviral therapy as indicated;
11. Patients with a history or current evidence of any concomitant condition, therapy, or laboratory abnormality that, in the opinion of the Investigator, might confound the results of the trial, interfere with the patient's participation and compliance;
12. Women who are lactating or pregnant, as confirmed by pregnancy test within 7 days before first treatment;
13. Male and female subjects who are unwilling to use adequate contraceptive methods (e.g., concomitant use of a spermicidal agent, barrier contraceptive, or/and intrauterine contraceptive) during the study and for at least 7 months after the last dose of GQ1001.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs). | End of Cycle 1 (21-day cycle)
  Adverse events will be assessed using NCI CTCAE version 5.0 and will be evaluated by the investigator and the sponsor for the eligibility of DLT.
Maximum Tolerated Dose (MTD) or Dose Recommended for Dose Expansion (DRDE) | After each cohort completes the DLT observation period (Day 1 to Day 21 after the first dose of study treatment) or has a DLT or becomes not DLT-evaluable
  The SRC will also determine the MTD/DRDE based on the totality of data for all tested dose levels.

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) | from baseline to 30 days after last dose
  Safety and Tolerability of GQ1001
Number of Participants with Abnormal Laboratory Values | rom baseline through Cycle 8 (each cycle is 21 days) and up to 30 days from treatment discontinuationafter last dose
  Safety and Tolerability of GQ1001
Area Under the Plasma Concentration Versus Time Curve (AUC) of GQ1001 | through study completion, an average of 1 year
Peak Plasma Concentration of GQ1001 (Cmax) | through study completion, an average of 1 year
Time at which the Cmax is Observed (Tmax) | through study completion, an average of 1 year
Half Life of GQ1001 (T1/2) | through study completion, an average of 1 year
Mean Residence Time of GQ1001 (MRT) | through study completion, an average of 1 year
Volume of Distribution of GQ1001 (Vd) | through study completion, an average of 1 year
Preliminary Efficacy of GQ1001 Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and CT of MRI scans | through study completion, an average of 1 year
Immunogenicity | through study completion, an average of 1 year
  Anti-GQ1001 antibody/anti-therapeutic antibody
Preliminary Efficacy | through study completion, an average of 1 year
  objective response rate (ORR)
Preliminary Efficacy | through study completion, an average of 1 year
  disease control rate (DCR)
Preliminary Efficacy | through study completion, an average of 1 year
  duration of response (DoR)
Preliminary Efficacy | through study completion, an average of 1 year
  progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Locations (24):
- M.D. Anderson Cancer Center, Houston, Texas, United States
- Australia (2):
  - Scientia Clinical Research Limited, Randwick, New South Wales
  - Cabrini Institute in Melbourne, Australia, Melbourne, Victoria
- China (21):
  - The first affiliated hospital of Bengbu medical college, Bengbu, Anhui
  - Beijing Tongren Hospital Affiliated to Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA general hospital, Beijing, Beijing Municipality
  - Southern Medical University Hospital in the south, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Huazhong University of Science and provincial Cancer Hospital Affiliated Union Hospital of Tongji Medical College, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shandong Tumor Hospital, Jinan, Shandong
  - Shanghai Ninth People's Hospital affiliated with the Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China School of Medicine and West China Hospital, Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Zhou C, Wang B, Teng C, Yang H, Piha-Paul SA, Richardson G, Malalasekera A, Sun Y, Wang W, Liu J, Shi Y, Zhan X, Lemech C. A phase Ia study of a novel anti-HER2 antibody-drug conjugate GQ1001 in patients with previously treated HER2 positive advanced solid tumors. J Transl Med. 2025 Jan 9;23(1):37. doi: 10.1186/s12967-024-05985-z. PMID 39789619